CLINICAL TRIAL: NCT00511368
Title: Phase 2 Dose-escalating, P-C, D-B, Parallel Group Study in HIV Treatment-experienced Patients to Evaluate the Safety, Tolerability and Efficacy of PA103001-04 Administered as Functional Monotherapy for 14 Days *(PART B)
Brief Title: Phase 2 Safety and Efficacy Study of Bevirimat Functional Monotherapy in HIV Treatment-Experienced Patients for 2 Weeks*
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew Beelen, M.D, Sr. Director Clinical Research, Myriad Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PA103001-04 Study 203
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV; treatment experienced; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — bevirimat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): placebo
  Interventions: Drug: matching placebo
- 2 (Experimental): Bevirimat
  Interventions: Drug: matching placebo; Drug: Bevirimat

INTERVENTIONS:
Drug: matching placebo
  Other Names: PA103001-04; PA-457N
Drug: Bevirimat
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate antiretroviral activity of up to five different oral doses administered for two weeks of bevirimat versus placebo in HIV treatment experienced patients, who have documented genotypic resistance to at least one major mutation from the IAS-USA list (2007)of resistance mutations for NRTIs, NNRTIs, or PIs. Patients will also be monitored for side effects, and the pharmacokinetics of bevirimat will be determined.

DETAILED DESCRIPTION:
Bevirimat (PA103001-04) represents a new class of antivirals that blocks HIV replication by disrupting virus maturation; specifically, by inhibiting a late step in the Gag processing cascade. Short term (7-10 days) functional monotherapy studies (conducted in patients with detectable viral loads on a failing regimen)help in determining the potency of the drug, and enable dose finding. This is a two part (A and B)randomized, placebo-controlled, double-blind, multiple-dose, dose-escalation study in HIV treatment-experienced patients on a failing regimen (harboring resistance mutations to at least one member of the NRTI, NNRTI or PI classes. The antiretroviral activity, safety, and pharmacokinetics of up to 5 different dose levels of bevirimat will be compared to placebo when added to a failing approved antiretroviral regimen. The study is conducted in two parts: A and B. In Part A following 14 days of daily dosing patients commenced a new optimized ART regimen in addition to their randomized treatment. In Part Part B dosing with the randomized treatment ends after the initial 14 days of daily dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Females of child-bearing potential, must have a documented negative pregnancy test and be willing to utilize double-barrier contraception through-out the study period.
* Have HIV-1-infection.
* Have a screening plasma HIV-1 RNA value, measured by the Roche Amplicor assay, of 2,000 - 250,000 copies/ml (inclusive).
* Have documented evidence of genotypic resistance in their medical records (at screening) or have resistance at screening by genotype to any major mutation from the IAS-USA list of resistance drug mutations, defined as: NRTI resistance: M41L, K65R, D67N, K70R, K70E, L74V, Y115F, M184V, M184V/I, L210W, T215Y/F, K219Q/E; NNRTI resistance: L100I, K103N, V106M, V106A/M, V108I, Y181C, Y181C/I, Y188L, Y188C/L/H, G190S/A, G190A, P225H; Major PI resistance: D30N, V32I, L33F, M46I/L, I47V/A, G48V, I50L, I50V, I54M/L, L76V, V82A/F/T, V82A/F/T/S, V82L/T, I84V, N88S, L90M
* Be receiving an antiretroviral therapy regimen containing at least 3 drugs (regimens containing ritonavir must not exceed a total daily dose of 400 mg) which has been unchanged for at least 8 weeks prior to initial screening.
* Be able to receive an optimized background regimen.
* Be free from any acute infection or serious medical illness within 14 days prior to study entry.
* Be informed of the nature of the study and provide written informed consent.
* Be willing to comply with the meal requirements described in the protocol.

Exclusion Criteria:

* Current opportunistic infection characteristic of AIDS
* Patients unable or unwilling to comply with the dosing schedule and protocol evaluations.
* Patients with malabsorption syndromes affecting drug absorption.
* Patients with systolic blood pressure < 90 mmHg or > 140 mmHg or diastolic blood pressure < 60 mmHg or > 90 mmHg measured in a semi-recumbent position after at least 10 minutes of rest at the screening or qualification visit.
* A history of seizures (excluding pediatric febrile seizures), migraines, cluster and/or chronic headaches, cerebrovascular accident (CVA) or transient ischemic attacks (TIA).
* Patients with abnormal Hemoglobin (< 10.0 g/dL for men and < 9.0 g/dL for women), Neutrophil count (< 1000/mm3), Platelet count (< 100,000/mm3), AST or ALT > 2.5 times the upper limit of normal (patients with a positive HBV surface antigen or HCV antibody test at screening must have AST and ALT no more than 1.5 times the upper limit of normal)
* Patients who have received radiation therapy or cytotoxic chemotherapeutic agents, immunomodulating agents, HIV immunotherapeutic vaccine, an investigational drug or product, or participation in a drug study within 4 weeks prior to the first dose of study drug.
* A history of alcoholism or drug addiction within the past 1 year (unless enrolled in a treatment program and approved by the sponsor). Recent use of any recreational drugs (except marijuana).
* A history of difficulty donating blood or inadequate venous access.
* The donation of blood or plasma within 30 days prior to receiving study medication.

Note: patients with a CD4 count <100 cells/mm3 will be considered for enrollment following discussion and agreement between the Investigator and the Sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA change from baseline over the first 14 days of study | 14 days

SECONDARY OUTCOMES:
safety and tolerability; pharmacokinetics | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, M.D., Study Director — Myrexis Inc.
Locations (18):
- United States (18):
  - UCLA Medical Center, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado Health Science Center, Denver, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Gary Richmond, Fort Lauderdale, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AIDS Research Consortium of Atlanta, Inc., Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The Research Insitute, Boston, Massachusetts
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Miriam Hospital/Brown University, Providence, Rhode Island
  - Central Texas Clinical Research, Austin, Texas
  - Southwest Infectious Diseases, Dallas, Texas
  - University of Texas Medical Branch Internal Medicine, Galveston, Texas

REFERENCES:
- See also: Related Info — http://www.hivforum.org
- See also: Related Info — http://www.amfar.org
- See also: Related Info — http://www.hivandhepatitis.com
- See also: Related Info — http://www.medscape.com